CLINICAL TRIAL: NCT02060344
Title: Hispanic Community Health Study / Study of Latinos (HCHS/SOL)
Brief Title: Hispanic Community Health Study / Study of Latinos
Acronym: HCHS/SOL
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HCHS-SOL; HHSN268201300001I (Other Grant/Funding Number: NHLBI); HHSN268201300002I (Other Grant/Funding Number: NHLBI); HHSN268201300003I (Other Grant/Funding Number: NHLBI); HHSN268201300004I (Other Grant/Funding Number: NHLBI); HHSN268201300005I (Other Grant/Funding Number: NHLBI); HHSN268201300024C (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2014-01-31; First posted 2014-02-12 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Hispanic; Latinos
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and DNA samples were collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hispanic/Latinos residing in the US: The cohort consists of over 16,400 persons of Hispanic/Latino origin, ages 18-74, specifically Cuban, Puerto Rican, Mexican, and Central/South American, to be recruited through four Field Centers affiliated with San Diego State University, Northwestern University in Chicago, Albert Einstein College of Medicine in the Bronx area of New York, and the University of Miami.

SUMMARY:
The Hispanic Community Health Study / Study of Latinos (HCHS/SOL) is a multi-center epidemiologic study in Hispanic/Latino populations to determine the role of acculturation in the prevalence and development of disease, and to identify risk factors playing a protective or harmful role in Hispanics/Latinos.

DETAILED DESCRIPTION:
Study goals include studying the prevalence and development of disease in Hispanics/Latinos, the role of acculturation, and to identify risk factors that play protective or harmful roles in Hispanics/Latinos. The target population of 16,000 persons of Hispanic/Latino origin, specifically Cuban, Puerto Rican, Mexican, and Central/South American, to be recruited through four Field Centers affiliated with San Diego State University, Northwestern University in Chicago, Albert Einstein College of Medicine in the Bronx area of New York, and the University of Miami. Seven additional academic centers serve as scientific and logistical support centers.

Study participants aged 18-74 years underwent an extensive clinic exam and assessments to determine baseline risk factors. Annual follow-up interviews will be conducted for 2-4 years to determine health outcomes of interest. Study results will be disseminated through scientific journals and also conveyed to the communities involved in the study in order to improve public health at the local level. Annual follow-up interviews will be conducted for 2-4 years to determine health outcomes of interest. Study results will be disseminated through scientific journals and also conveyed to the communities involved in the study in order to improve public health at the local level.

ELIGIBILITY:
Inclusion Criteria:

• Hispanic/Latino persons living in the US, aged 18-74 in four communities: San Diego, Bronx NY, Chicago, and Miami.Examination of the cohort following a standardized protocol

Exclusion Criteria:

* Plans to move from the region within 6 months.
* Unable to complete the study questionnaires in English or Spanish.
* Women who are pregnant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The of over 16,400 persons of Hispanic/Latino origin, specifically Cuban, Puerto Rican, Mexican, and Central/South American, to be recruited through four Field Centers affiliated with San Diego State University, Northwestern University in Chicago, Albert Einstein College of Medicine in the Bronx area of New York, and the University of Miami.
Sampling Method: Probability Sample
Enrollment: 16400 (Actual)
Dates: Start 2006-01; Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiovascular and pulmonary disease risk factors in Hispanics/Latinos | Visit 2 data collection through 2019, preliminary and final analyses through 2019, Annual Follow-up through 2019
  This is a population-based cohort study of 16,400 Hispanic/Latinos. Objectives:
  * Examination of the cohort following a standardized protocol
  * Follow-up of the cohort to assess vital status, changes in health status, medication intake, and new cardiovascular and pulmonary events (fatal and non-fatal MI, heart failure, stroke, asthma, and COPD.
  * Understand the relationship between changes in risk factors and protective factors and onset of CV and pulmonary disease progression
  * Understand the relationship between changes in sociocultural factors and changes in health
  * Understand the relationship between baseline CV risk profile of women of childbearing age and incidence of select pregnancy complications

CONTACTS AND LOCATIONS:
Overall Officials: Jianwen Cai, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Robert Kaplan, PhD, Principal Investigator — Einstein College of Medicine; Neil Schneiderman, PhD, Principal Investigator — University of Miami; Gregory Talavera, MD, MPH, Principal Investigator — San Diego State University; Martha Daviglus, MD, PhD, Principal Investigator — University of Illinois at Chicago; Scott Solomon, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Sorlie PD, Aviles-Santa LM, Wassertheil-Smoller S, Kaplan RC, Daviglus ML, Giachello AL, Schneiderman N, Raij L, Talavera G, Allison M, Lavange L, Chambless LE, Heiss G. Design and implementation of the Hispanic Community Health Study/Study of Latinos. Ann Epidemiol. 2010 Aug;20(8):629-41. doi: 10.1016/j.annepidem.2010.03.015. PMID 20609343
- [Derived] Isasi CR, Gallo LC, Cai J, Gellman MD, Xie W, Heiss G, Kaplan RC, Talavera GA, Daviglus ML, Pirzada A, Wassertheil-Smoller S, Llabre MM, Youngblood ME, Schneiderman N, Perez-Stable EJ, Napoles AM, Perreira KM. Economic and Psychosocial Impact of COVID-19 in the Hispanic Community Health Study/Study of Latinos. Health Equity. 2023 Mar 27;7(1):206-215. doi: 10.1089/heq.2022.0211. eCollection 2023. PMID 37007686
- [Derived] Alvarez CS, Aviles-Santa ML, Freedman ND, Perreira KM, Garcia-Bedoya O, Kaplan RC, Daviglus ML, Graubard BI, Talavera GA, Thyagarajan B, Camargo MC. Associations of Helicobacter pylori and hepatitis A seropositivity with asthma in the Hispanic Community Health Study/Study of Latinos (HCHS/SOL): addressing the hygiene hypothesis. Allergy Asthma Clin Immunol. 2021 Nov 24;17(1):120. doi: 10.1186/s13223-021-00625-3. PMID 34819160
- [Derived] Maldonado LE, Adair LS, Sotres-Alvarez D, Mattei J, Mossavar-Rahmani Y, Perreira KM, Daviglus ML, Van Horn LV, Gallo LC, Isasi CR, Albrecht SS. Dietary Patterns and Years Living in the United States by Hispanic/Latino Heritage in the Hispanic Community Health Study/Study of Latinos (HCHS/SOL). J Nutr. 2021 Sep 4;151(9):2749-2759. doi: 10.1093/jn/nxab165. PMID 34320207
- [Derived] Bai F, Chen J, Pandey D, Durazo-Arvizu R, Talavera GA, Allison MA, Perreira KM, Schneiderman N, Sutherland MW, Cai J, Daviglus ML, Testai FD. Stroke Risk Factor Status and Use of Stroke Prevention Medications Among Hispanic/Latino Adults in HCHS/SOL. Stroke. 2021 Apr;52(4):1339-1346. doi: 10.1161/STROKEAHA.120.031216. Epub 2021 Mar 4. PMID 33657859
- [Derived] Chen GC, Qi Q, Hua S, Moon JY, Spartano NL, Vasan RS, Sotres-Alvarez D, Castaneda SF, Evenson KR, Perreira KM, Gallo LC, Pirzada A, Diaz KM, Daviglus ML, Gellman MD, Kaplan RC, Xue X, Mossavar-Rahmani Y. Accelerometer-assessed physical activity and incident diabetes in a population covering the adult life span: the Hispanic Community Health Study/Study of Latinos. Am J Clin Nutr. 2020 Nov 11;112(5):1318-1327. doi: 10.1093/ajcn/nqaa232. PMID 32910816
- [Derived] Chen GC, Chai JC, Yu B, Michelotti GA, Grove ML, Fretts AM, Daviglus ML, Garcia-Bedoya OL, Thyagarajan B, Schneiderman N, Cai J, Kaplan RC, Boerwinkle E, Qi Q. Serum sphingolipids and incident diabetes in a US population with high diabetes burden: the Hispanic Community Health Study/Study of Latinos (HCHS/SOL). Am J Clin Nutr. 2020 Jul 1;112(1):57-65. doi: 10.1093/ajcn/nqaa114. PMID 32469399
- [Derived] Elfassy T, Mossavar-Rahmani Y, Van Horn L, Gellman M, Sotres-Alvarez D, Schneiderman N, Daviglus M, Beasley JM, Llabre MM, Shaw PA, Prado G, Florez H, Zeki Al Hazzouri A. Associations of Sodium and Potassium with Obesity Measures Among Diverse US Hispanic/Latino Adults: Results from the Hispanic Community Health Study/Study of Latinos. Obesity (Silver Spring). 2018 Feb;26(2):442-450. doi: 10.1002/oby.22089. Epub 2018 Jan 10. PMID 29318759
- [Derived] Corsino L, Sotres-Alvarez D, Butera NM, Siega-Riz AM, Palacios C, Perez CM, Albrecht SS, Espinoza Giacinto RA, Perera MJ, Horn LV, Aviles-Santa ML. Association of the DASH dietary pattern with insulin resistance and diabetes in US Hispanic/Latino adults: results from the Hispanic Community Health Study/Study of Latinos (HCHS/SOL). BMJ Open Diabetes Res Care. 2017 Jul 7;5(1):e000402. doi: 10.1136/bmjdrc-2017-000402. eCollection 2017. PMID 28761660
- [Derived] Mattei J, Sotres-Alvarez D, Daviglus ML, Gallo LC, Gellman M, Hu FB, Tucker KL, Willett WC, Siega-Riz AM, Van Horn L, Kaplan RC. Diet Quality and Its Association with Cardiometabolic Risk Factors Vary by Hispanic and Latino Ethnic Background in the Hispanic Community Health Study/Study of Latinos. J Nutr. 2016 Oct;146(10):2035-2044. doi: 10.3945/jn.116.231209. Epub 2016 Sep 7. PMID 27605403
- [Derived] Wong WW, Strizich G, Heo M, Heymsfield SB, Himes JH, Rock CL, Gellman MD, Siega-Riz AM, Sotres-Alvarez D, Davis SM, Arredondo EM, Van Horn L, Wylie-Rosett J, Sanchez-Johnsen L, Kaplan RC, Mossavar-Rahmani Y. Relationship between body fat and BMI in a US hispanic population-based cohort study: Results from HCHS/SOL. Obesity (Silver Spring). 2016 Jul;24(7):1561-71. doi: 10.1002/oby.21495. Epub 2016 May 17. PMID 27184359
- [Derived] Oelsner EC, Loehr LR, Henderson AG, Donohue KM, Enright PL, Kalhan R, Lo Cascio CM, Ries A, Shah N, Smith BM, Rosamond WD, Barr RG. Classifying Chronic Lower Respiratory Disease Events in Epidemiologic Cohort Studies. Ann Am Thorac Soc. 2016 Jul;13(7):1057-66. doi: 10.1513/AnnalsATS.201601-063OC. PMID 27088163
- [Derived] Mossavar-Rahmani Y, Jung M, Patel SR, Sotres-Alvarez D, Arens R, Ramos A, Redline S, Rock CL, Van Horn L. Eating behavior by sleep duration in the Hispanic Community Health Study/Study of Latinos. Appetite. 2015 Dec;95:275-84. doi: 10.1016/j.appet.2015.07.014. Epub 2015 Jul 16. PMID 26189885
- [Derived] Mossavar-Rahmani Y, Shaw PA, Wong WW, Sotres-Alvarez D, Gellman MD, Van Horn L, Stoutenberg M, Daviglus ML, Wylie-Rosett J, Siega-Riz AM, Ou FS, Prentice RL. Applying Recovery Biomarkers to Calibrate Self-Report Measures of Energy and Protein in the Hispanic Community Health Study/Study of Latinos. Am J Epidemiol. 2015 Jun 15;181(12):996-1007. doi: 10.1093/aje/kwu468. Epub 2015 May 20. PMID 25995289
- [Derived] Siega-Riz AM, Sotres-Alvarez D, Ayala GX, Ginsberg M, Himes JH, Liu K, Loria CM, Mossavar-Rahmani Y, Rock CL, Rodriguez B, Gellman MD, Van Horn L. Food-group and nutrient-density intakes by Hispanic and Latino backgrounds in the Hispanic Community Health Study/Study of Latinos. Am J Clin Nutr. 2014 Jun;99(6):1487-98. doi: 10.3945/ajcn.113.082685. Epub 2014 Apr 23. PMID 24760972
- See also: HCHS/SOL — https://sites.cscc.unc.edu/hchs/
- Available data/document: Individual Participant Data Set: HCHS-SOL — http://biolincc.nhlbi.nih.gov/studies/hchssol/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/hchssol/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/hchssol/